CLINICAL TRIAL: NCT04422457
Title: Specific Molecular Imaging of DX600 Labeled by PET Radionuclide Targeting ACE2 in Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020KT62
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging cohort (Experimental): All study participants will be allocated to this arm (single-arm study).Study participants will undergo 68Ga-DX600 PET/CT scans
  Interventions: Other: 68Ga-DX600 PET/CT

INTERVENTIONS:
Other: 68Ga-DX600 PET/CT — DX600, labeled with 68Ga will be used as a molecular imaging tracer for PET/CT scanning

SUMMARY:
Angiotensin-converting enzyme 2 (ACE2) plays an important role in renin-angiotensin system (RAS) and has been reported to relate with cancer. Recently, it has also been proved as the key target for COVID-19 infection.

DX600 is a polypeptide that can specific binding to ACE2 specifically with nanomolar affinity reported in literature. This study constrcuted a radio-tracer, DX600 Labeled by PET Radionuclide, to monitoring biodistribution ACE2 in human beings, evaluate the detection ability of radio-tracer in ACE2 over-expression tumors and dynamic changes of ACE2 expression under therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old; both sex;
* ECoG 0 or 1;
* Patients that would undergo biopsy or surgical operation with high ACE2 expression tumors such as colorectal cancer, renal cancer, pancreatic cancer, gastric cancer, liver cancer, lung cancer, brain cancer or suspected tumor.
* use 18F-FDG PET/CT as baseline evaluation

Exclusion Criteria:

* Significant hepatic or renal dysfunction;
* Is Pregnant or ready to pregnant;
* Cannot lie on their back for half an hour;
* Suffering from claustrophobia or other mental diseases;
* Refusal to join the clinical study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
SUV | 2 years
  The uptake of uptake of the tracer in the primary and metastatic tumor lesions by measuring standardized uptake value（SUV）

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Q, Liu T, Ding J, Zhou N, Yu Z, Ren Y, Qin X, Du P, Yang Z, Zhu H. Evaluation of 68Ga- and 177Lu-Labeled HZ20 Angiotensin-Converting Enzyme 2-Targeting Peptides for Tumor-Specific Imaging. Mol Pharm. 2022 Nov 7;19(11):4149-4156. doi: 10.1021/acs.molpharmaceut.2c00541. Epub 2022 Oct 5. PMID 36198565